CLINICAL TRIAL: NCT01169519
Title: Safety, Pharmacokinetics and Hemodynamic Efficacy of Sildenafil in Single Ventricle Patients
Brief Title: Sildenafil in Single Ventricle Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00025220
Record Dates: First submitted 2010-07-07; First posted 2010-07-26 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2012-11

CONDITIONS: Heart Disease
Keywords: Hypoplastic left heart syndrome; Hypoplastic right heart syndrome; Superior cavopulmonary anastomosis; Total cavopulmonary anastomosis; Children with single ventricle anatomy
MeSH Terms: conditions — Heart Diseases; Hypoplastic Left Heart Syndrome | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sildenafil (Active Comparator): Pharmacokinetic and hemodynamic evaluation following sildenafil administration
  Interventions: Drug: Sildenafil by injection

INTERVENTIONS:
Drug: Sildenafil by injection — Sildenafil 0.125mg/kg injection over 20min
  Other Names: Revatio
Drug: Sildenafil by injection — Sildenafil 0.25mg/kg injection over 20min
  Other Names: Revatio
Drug: Sildenafil by injection — Sildenafil 0.35mg/kg by injection over 20min
  Other Names: Revatio
Drug: Sildenafil by injection — Sildenafil 0.45mg/kg by injection over 20min
  Other Names: Revatio

SUMMARY:
Patients with single ventricle anatomy undergo staged surgical palliation. The result is an "in series" circulation with pulmonary blood flow and cardiac output directly related to pulmonary vascular resistance. While surgical outcomes have improved, the physiology of the single ventricle palliation results in continued long term attrition. Elevated pulmonary vascular resistance and impaired systemic ventricular function are important risk factors for failure of single ventricle palliation.

Sildenafil is a pulmonary vasodilator and has been shown to improve cardiac contractility in the pressure overloaded right ventricle.

The investigators will assess the safety, pharmacokinetics and hemodynamic efficacy of sildenafil in single ventricle patients following stage II and III surgical palliation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 3 months; ≤120 months.
2. History of congenital heart disease with severe hypoplasia of a right or left ventricle.
3. Undergoing cardiac catheterization as part of standard clinical care.
4. Availability and willingness of the parent/legally authorized representative to provide written informed consent.

Exclusion Criteria:

1. History of serious adverse event related to sildenafil administration.
2. History of sildenafil exposure within 48 hours of the study.
3. Presence of pulmonary venous obstruction.
4. Treatment with organic nitrates or alpha blockade therapy.
5. Contraindication to cardiac catheterization as determined by the attending cardiologist and including:

   1. Significant hemodynamic instability.
   2. Sepsis.
   3. Need for Extra-Corporeal Membrane Oxygenation (ECMO) support.
   4. Venous occlusion precluding adequate access.
   5. Recent systemic illness.
6. Renal failure defined as serum creatinine > 2 times higher than the upper limit of normal.
7. Liver dysfunction defined as alanine aminotransferase or aspartate aminotransferase > 3 times higher than the upper limit of normal.
8. Thrombocytopenia defined as a platelet count < 50 000 cells/µL.
9. Leukopenia defined as white blood cells < 2500 cells/µL.

Ages: 3 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Hill, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Hill KD, Tunks RD, Barker PC, Benjamin DK Jr, Cohen-Wolkowiez M, Fleming GA, Laughon M, Li JS. Sildenafil exposure and hemodynamic effect after stage II single-ventricle surgery. Pediatr Crit Care Med. 2013 Jul;14(6):593-600. doi: 10.1097/PCC.0b013e31828aa5ee. PMID 23823195
- [Derived] Tunks RD, Barker PC, Benjamin DK Jr, Cohen-Wolkowiez M, Fleming GA, Laughon M, Li JS, Hill KD. Sildenafil exposure and hemodynamic effect after Fontan surgery. Pediatr Crit Care Med. 2014 Jan;15(1):28-34. doi: 10.1097/PCC.0000000000000007. PMID 24201857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited upon presentation for elective Pre-stage II or stage III catheterization. The first patient was recruited on 4/14/2011 and the final patient was enrolled on 11/29/2012
Pre-assignment Details: Enrolled subjects were excluded from trial participation if they demonstrated baseline hemodynamics suggesting that they would not tolerate sildenafil infusion (e.g. baseline hypotension)
Groups:
- Baseline/Sildenafil: Assessment of baseline hemodynamics followed by sildenafil infusion with repeat assessment of hemodynamics
Period: Overall Study
Arm/Group | Baseline/Sildenafil
Started | 21 (This was a pre-post study, All patients receiving a baseline assessment, also received sildenafil.)
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Overall 21 subjects were enrolled and all subjects received a baseline assessment followed by sildenafil administration.
Groups:
- Sildenafil: Pharmacokinetic and hemodynamic evaluation following sildenafil administration
  Sildenafil by injection : Sildenafil 0.45mg/kg by injection over 20min
  Sildenafil by injection : Sildenafil 0.25mg/kg injection over 20min
  Sildenafil by injection : Sildenafil 0.35mg/kg by injection over 20min
  Sildenafil by injection : Sildenafil 0.125mg/kg injection over 20min
Arm/Group | Sildenafil
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 3.4 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Sildenafil Plasma Concentration
Description: Assessment of peak sildenafil plasma concentration.
Time Frame: 5 minutes after completion of sildenafil infusion
Population: 3 patients were enrolled in this group but in 1 participant, an inadequate plasma sample volume prevented accurate determination of sildenafil concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Peak Sildenafil Level (ng/mL) for Dose = 0.125mg/kg; Peak Sildenafil Level (ng/mL) for Dose = 0.35mg/kg; Peak Sildenafil Level (ng/mL) for Dose = 0.45mg/kg: Maximum sildenafil plasma concentration measured 5 minutes after completion of sildenafil infusion
- Peak Sildenafil Level (ng/mL) for Dose = 0.25mg/kg: Maximum sildenafil plasma concentration measured 5 minutes after completion of sildenafil infusionplasma concentration
Arm/Group | Peak Sildenafil Level (ng/mL) for Dose = 0.125mg/kg | Peak Sildenafil Level (ng/mL) for Dose = 0.35mg/kg | Peak Sildenafil Level (ng/mL) for Dose = 0.45mg/kg | Peak Sildenafil Level (ng/mL) for Dose = 0.25mg/kg
Number analyzed (Participants) | 2 | 8 | 5 | 5
ng/mL | 181 (126) | 515 (98) | 545 (185) | 202 (92)

2. Secondary Outcome: Hemodynamic Safety and Efficacy
Description: Assessment of pulmonary vascular resistance
Time Frame: 10 minutes after completion of sildenafil infusion
Measure: Median (Inter-Quartile Range); unit: Wood units * m^2
Groups:
- Baseline: Assessment of baseline hemodynamics
Arm/Group | Baseline | Sildenafil
Number analyzed (Participants) | 21 | 21
Wood units * m^2 | 2.3 [1.7 to 3.0] | 1.6 [1.2 to 2.0]

ADVERSE EVENTS:
Groups:
- Dose = 0.125mg/kg: Subjects receiving a sildenafil dose of 0.125mg/kg IV over 20 min
- Dose = 0.25mg/kg: Subjects receiving a sildenafil dose of 0.25mg/kg IV over 20 min
- Dose = 0.35mg/kg: Subjects receiving a sildenafil dose of 0.35mg/kg IV over 20 min
- Dose = 0.45mg/kg: Subjects receiving a sildenafil dose of 0.45mg/kg IV over 20 min
Arm/Group | Dose = 0.125mg/kg | Dose = 0.25mg/kg | Dose = 0.35mg/kg | Dose = 0.45mg/kg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/8 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No